CLINICAL TRIAL: NCT02934347
Title: Comparison of Glottic Views and Intubation Times in the Supine and 25 Degree Back-up Positions
Status: Completed | Type: Observational
Sponsor: Betsi Cadwaladr University Health Board (Other Government)
Responsible Party: Principal Investigator, Raj M Reddy, Consultant Anaesthetist, Betsi Cadwaladr University Health Board
Other Study IDs: BetsiCUHB
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-04

CONDITIONS: Elective Surgical Patients
Keywords: Intubation, Back-up position; Glottis, View

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Supine: A baseline group of adult patients who required intubation as part of their routine anaesthesia who were intubated in the standard horizontal sniffing position.
- Back-up: A subsequent group of similar the patients who had their anaesthesia induced and tracheas intubated in a 25 degree back-up position achieved by flexion of the operating table at the hips
  Interventions: Procedure: 25 degree back-up position

INTERVENTIONS:
Procedure: 25 degree back-up position — To test whether a 25 degree back-up position improves laryngeal views and makes intubation easier compared to the standard horizontal position
  Groups: Back-up

SUMMARY:
Our hypothesis is that the view of the glottis may be improved by putting all patients requiring intubation in the ramped or back up position while maintaining the classic sniffing position.

DETAILED DESCRIPTION:
The sniffing position has traditionally been considered the optimal head position for direct laryngoscopy and is the usual patient position preferred by most anaesthetists. In theory, neck flexion aligns the pharyngeal and laryngeal axes, and head extension at the atlanto-occipital joint aligns the oral axis with these two axes allowing the line of sight to fall on the glottis. It is recognized as the starting head position for direct laryngoscopy because it provides the best chance of adequate exposure.

However the sniffing position does not guarantee adequate exposure in all patients because many other anatomical factors control the final degree of visualization.

To achieve a proper sniffing position in obese patients, the "ramped" (or the back-up) position has been used as this produces better neck flexion and head extension in these patients when compared to the horizontal supine position. Also the forces required to elevate and move the tongue and other tissues out of the line of sight are less when the patients are ramped.

Our hypothesis is that the view of the glottis may be improved by putting all (ie not only obese) patients requiring intubation in the ramped or back up position while maintaining the classic sniffing position.

ELIGIBILITY:
Inclusion Criteria:

* Adult surgical patients who required intubation as part of their routine anaesthesia

Exclusion Criteria:

1. Patients less than 18 years old,
2. Patients recognised to have difficult airways where an alternative method of intubation (e.g. fibre optic) was the method of choice,
3. Patients undergoing emergency surgery where patient positioning and data collection might cause delay (e.g. exsanguinating patients) or where the supine position is not optimal (e.g. brisk bleeding into the upper airway),
4. Patients requiring rapid sequence induction of anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who required intubation as part of their routine anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 781 (Actual)
Dates: Start 2012-02; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raj M Reddy, FRCA, Principal Investigator — Anaesthetic Department, Glan Clwyd Hospital, Betsi Cadwaladr University Health Board

IPD SHARING:
Plan to Share IPD: Yes
Publish anonymised raw data as supplementary file

REFERENCES:
- [Background] Adnet F, Baillard C, Borron SW, Denantes C, Lefebvre L, Galinski M, Martinez C, Cupa M, Lapostolle F. Randomized study comparing the "sniffing position" with simple head extension for laryngoscopic view in elective surgery patients. Anesthesiology. 2001 Oct;95(4):836-41. doi: 10.1097/00000542-200110000-00009. PMID 11605921
- [Background] Bannister FB, Macbeth RG. Direct laryngoscopy and tracheal intubation. Lancet 1944; 2: 651-4
- [Background] Greenland KB, Edwards MJ, Hutton NJ, Challis VJ, Irwin MG, Sleigh JW. Changes in airway configuration with different head and neck positions using magnetic resonance imaging of normal airways: a new concept with possible clinical applications. Br J Anaesth. 2010 Nov;105(5):683-90. doi: 10.1093/bja/aeq239. Epub 2010 Sep 15. PMID 20846964
- [Background] Jackson C. Bronchoscopy and Esophagoscopy: A Manual of Peroral Endoscopy and Laryngeal Surgery. Philadelphia and London: WB Saunders; 1922
- [Background] Lee BJ, Kang JM, Kim DO. Laryngeal exposure during laryngoscopy is better in the 25 degrees back-up position than in the supine position. Br J Anaesth. 2007 Oct;99(4):581-6. doi: 10.1093/bja/aem095. Epub 2007 Jul 4. PMID 17611252
- [Background] Lee HC, Yun MJ, Hwang JW, Na HS, Kim DH, Park JY. Higher operating tables provide better laryngeal views for tracheal intubation. Br J Anaesth. 2014 Apr;112(4):749-55. doi: 10.1093/bja/aet428. Epub 2013 Dec 18. PMID 24355831
- [Background] Rao SL, Kunselman AR, Schuler HG, DesHarnais S. Laryngoscopy and tracheal intubation in the head-elevated position in obese patients: a randomized, controlled, equivalence trial. Anesth Analg. 2008 Dec;107(6):1912-8. doi: 10.1213/ane.0b013e31818556ed. PMID 19020138
- [Background] Collins JS, Lemmens HJ, Brodsky JB, Brock-Utne JG, Levitan RM. Laryngoscopy and morbid obesity: a comparison of the "sniff" and "ramped" positions. Obes Surg. 2004 Oct;14(9):1171-5. doi: 10.1381/0960892042386869. PMID 15527629
- [Background] Lane S, Saunders D, Schofield A, Padmanabhan R, Hildreth A, Laws D. A prospective, randomised controlled trial comparing the efficacy of pre-oxygenation in the 20 degrees head-up vs supine position. Anaesthesia. 2005 Nov;60(11):1064-7. doi: 10.1111/j.1365-2044.2005.04374.x. PMID 16229689
- [Background] Dixon BJ, Dixon JB, Carden JR, Burn AJ, Schachter LM, Playfair JM, Laurie CP, O'Brien PE. Preoxygenation is more effective in the 25 degrees head-up position than in the supine position in severely obese patients: a randomized controlled study. Anesthesiology. 2005 Jun;102(6):1110-5; discussion 5A. doi: 10.1097/00000542-200506000-00009. PMID 15915022
- [Background] Lebowitz PW, Shay H, Straker T, Rubin D, Bodner S. Shoulder and head elevation improves laryngoscopic view for tracheal intubation in nonobese as well as obese individuals. J Clin Anesth. 2012 Mar;24(2):104-8. doi: 10.1016/j.jclinane.2011.06.015. Epub 2012 Feb 1. PMID 22301204
- [Derived] Reddy RM, Adke M, Patil P, Kosheleva I, Ridley S; Anaesthetic Department at Glan Clwyd Hospital. Comparison of glottic views and intubation times in the supine and 25 degree back-up positions. BMC Anesthesiol. 2016 Nov 16;16(1):113. doi: 10.1186/s12871-016-0280-4. PMID 27852241

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supine | Back-up
Started | 374 | 407
Completed | 374 | 407
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Supine | Back-up | Total
Number analyzed (Participants) | 374 | 407 | 781
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (17.6) | 55.8 (16.9) | 56.6 (17.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One patient's gender was not recorded
  Participants
    number analyzed (Participants) | 374 | 406 | 780
    Female | 188 | 218 | 406
    Male | 186 | 188 | 374
Region of Enrollment [Number; unit: participants]
  United Kingdom | 374 | 407 | 781
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 28.5 (5.5) | 28 (5.8) | 28.2 (5.6)
Type of surgery [Number; unit: participants]
  General | 248 | 233 | 481
  Gynaecology | 44 | 24 | 68
  Urology | 29 | 19 | 48
  ENT | 24 | 43 | 67
  Ophthalmology | 0 | 1 | 1
  Orthopaedics | 12 | 3 | 15
  Facio-Maxillary | 10 | 62 | 72
  Trauma | 4 | 18 | 22
  Vascular | 2 | 4 | 6
  Not recorded | 1 | 0 | 1
Grade of intubating anaesthetist [Number; unit: participants] — Senior anaesthetists were permanent fulled trained members of staff capable of independent practice.
  Trainee anaesthetists were on approved training programmes, required supervision by a nominated senior anaesthetist and rotated to Glan Clwyd Hospital for a fixed period of training.
  participants
    Senior | 272 | 264 | 536
    Not recorded | 1 | 0 | 1
    Trainee | 101 | 143 | 244

OUTCOME MEASURES:

1. Primary Outcome: The Best Glottic View Obtained During Laryngoscopy
Description: The best glottic view obtained during laryngoscopy was assessed using the Cormack and Lehane classification by the anaesthetist performing the laryngoscopy.
  The Cormack and Lehane classifies glottic views as follows: Grade 1: Most of the glottis is visible, Grade 2: At best almost half of the glottis is seen, at worst only the posterior tip of the arytenoids is seen., Grade 3: Only the epiglottis is visible, Grade 4: No laryngeal structures are visible.
Time Frame: The view of the glottis was measured once while the patient was being intubated
Population: Adult patients who required intubation as part of their routine anaesthesia
Measure: Number; unit: participants
Arm/Group | Supine | Back-up
Number analyzed (Participants) | 374 | 407
participants
  Cormack and Lehane Grade 1 | 186 | 228
  Cormack and Lehane Grade 2 | 163 | 151
  Cormack and Lehane Grade 3 | 23 | 24
  Cormack and Lehane Grade 4 | 2 | 2
  Not recorded | 0 | 2
Statistical Analysis 1: Comparison: Supine vs Back-up; Null hypothesis: no difference in frequency of grade of glottic view between the supine and back-up positions; Test type: Superiority or Other; p > 0.05, Chi-squared, Corrected — Grades analysed were 1, 2 and then 3 and 4 combined because of low frequencies in the latter two grades; Chi-squared for trend

2. Secondary Outcome: The Number of Attempts at Both Laryngoscopy and Tracheal Intubation
Description: The number of attempts at both laryngoscopy and tracheal intubation were recorded
Time Frame: Once at intubation
Population: Adult patients who required intubation as part of their routine anaesthesia
Measure: Number; unit: participants
Arm/Group | Supine | Back-up
Number analyzed (Participants) | 374 | 407
participants
  1 Laryngoscopy attempt | 340 | 371
  2 Laryngoscopy attempts | 25 | 27
  >2 Laryngoscopy attempts | 5 | 3
  Laryngoscopy attempts Not recorded | 4 | 6
  1 Intubation attempt | 346 | 378
  2 Intubation attempts | 22 | 18
  >2 Intubation attempts | 0 | 1
  Intubation attempts Not recorded | 6 | 10
Statistical Analysis 1: Comparison: Supine vs Back-up; Test type: Superiority or Other; p < 0.01, Chi-squared; df=3

3. Secondary Outcome: The Use of Ancillary Equipment
Description: The use of ancillary equipment (e.g. bougie, alternative laryngoscope blades) and manoeuvres (e.g. laryngeal manipulation) were recorded but applied at the intubating anaesthetist's discretion
Time Frame: Once at intubation
Population: Adult patients who required intubation as part of their routine anaesthesia
Measure: Number; unit: participants
Arm/Group | Supine | Back-up
Number analyzed (Participants) | 374 | 407
participants
  Ancillary equipment: Bougie | 58 | 61
  Other Ancillary equipment | 3 | 4
  Ancillary equipment: 'Not Used' | 308 | 341
  Ancillary equipment use not recorded | 5 | 1
  Ancillary manoeuvre: Cricoid | 19 | 2
  Ancillary manoeuvre: BURP | 34 | 25
  External laryngeal manipulation | 39 | 53
  Ancillary manoeuvres: 'Not Used' | 277 | 326
  Ancillary manoeuvres not recorded | 5 | 1
Statistical Analysis 1: Comparison: Supine vs Back-up; Test type: Superiority or Other; p > 0.05, Chi-squared

4. Secondary Outcome: The Time Between the Beginning of Laryngoscopy and Detection of Carbon Dioxide on the End-tidal Carbon Dioxide Monitor
Description: The time between the beginning of laryngoscopy and detection of carbon dioxide on the end-tidal carbon dioxide monitor after the successful placement of the tracheal tube was recorded
Time Frame: Once at intubation
Population: Adult patients who required intubation as part of their routine anaesthesia
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Supine | Back-up
Number analyzed (Participants) | 374 | 407
seconds
  Senior | 26 [17.25 to 40] | 21 [16 to 36]
  Trainee | 30 [22 to 47.50] | 27 [18.75 to 42]
  Senior & Trainee combined | 28 [18 to 42] | 24 [16 to 39]
Statistical Analysis 1: Comparison: Supine vs Back-up; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Any adverse events relating to assessing the glottic view were recorded. Such assessment occurred during intubation which took a minimum of 4 secs and an maximum of 7 mins 34 sec.
Arm/Group | Supine | Back-up
Serious Adverse Events (participants affected / at risk) | 0/374 | 0/407
Other Adverse Events (participants affected / at risk) | 0/374 | 0/407

LIMITATIONS AND CAVEATS:
The present study was under-powered to detect small differences in glottic views.

There would be additional variation as the results were reported by the whole Anaesthetic Dept rather than a few investigators

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes